CLINICAL TRIAL: NCT03227835
Title: Contrast-Induced Nephropathy After Revision of the Prophylaxis Threshold
Acronym: CINART
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2017-0058
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Contrast-induced Nephropathy
Keywords: contrast-induced nephropathy; contrast-induced acute kidney injury; prophylaxis; intravenous hydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intravascular iodinated contrast material administration — Evaluation of the consequences of the protocol change to not giving prophylaxis to patients with an eGFR >29mL/min/1.73m2

SUMMARY:
After administration of intravascular iodinated contrast media Contrast-Induced Nephropathy (CIN), also known as Contrast-Induced Acute Kidney Injury (CIAKI), may occur. CIN/CI-AKI is associated with increased risk of dialysis and mortality. No treatment exists for CIN/CI-AKI, therefore the focus lies on prevention. Clinical practice guidelines for the prevention of CIN/CI-AKI exist and are implemented in most hospitals. Generally, intravascular volume expansion with normal saline is recommended as prophylaxis.

Earlier this year the results of the AMACING study (A MAastricht Contrast-Induced Nephropathy Guideline study) were published in The Lancet (NL47173.068.14/METC 14-2-006; Clinical Trials.gov NCT02106234; http://www.thelancet.com/journals/lancet/article/PIIS0140-6736(17)30057-0/fulltext). These results show that for the greater part (>90%) of patients considered to be at risk of CIN/CI-AKI by the guidelines, withholding prophylaxis is non-inferior to giving standard intravenous prophylactic hydration in the prevention of CIN/CI-AKI. Furthermore, the standard prophylactic hydration confers some risk (5.5% complications of intravenous hydration were recorded in the AMACING study).

As a result the clinical protocol in the Maastricht University Medical Centre (MUMC+) has been adapted, and patients with an estimated Glomerular Filtration Rate (eGFR) >29mL/min/1.73m2 no longer receive intravenous prophylactic hydration before or after procedures with intravascular iodinated contrast material administration.

CINART is a one year prospective observational study with the aim to evaluate the consequences of the protocol change for 1. for incidences of CIN/CI-AKI, dialysis and mortality, 2. for clinical practice in terms of patient burden (complications of prophylaxis), hospital burden (extra hospitalisations for prophylaxis), and costs, as derived from the number of elective procedures carried out in patients formerly eligible for prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* referred for an elective procedure with intravascular iodinated contrast administration at Maastricht University Medical Centre
* eGFR30-44mL/min/1.73m2 OR eGFR45-59mL/min/1.73m2 + DM OR eGFR45-59mL/min/1.73m2 + >1 risk factor (>age >75 years, anaemia, cardiovascular disease, prescribed NSAID or Diuretic medication) OR multiple myeloma/lymphoplasmacytic lymphoma with small chain proteinuria.

Exclusion Criteria:

* eGFR<30mL/min/1.73m2
* Dialysis/renal replacement therapy
* emergency procedure
* intensive care patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk of CIN/CIAKI according to the guidelines and an eGFR between 30-59mL/min/1.73m2, who are referred for an elective procedure with intravascular iodinated contrast administration at the MUMC+ after the protocol change i.e. the threshold for prophylactic intravenous hydration has been lowered to eGFR<30mL/min/1.73m2.
Sampling Method: Non-Probability Sample
Enrollment: 1372 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of procedures | 1 year
  Number of elective procedures with intravascular contrast in patients formerly eligible for prophylaxis

SECONDARY OUTCOMES:
Contrast-Induced Nephropathy | 2-6 days post contrast administration
  >25% or >44umol/L increase in serum creatinine from baseline
1-month dialysis | 26-35 days post-contrast
  incidences of dialysis
1-month mortality | 26-35 days post-contrast
  incidences of all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: JE Wildberger, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Zuid-Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nijssen EC, Rennenberg RJ, Nelemans PJ, Essers BA, Janssen MM, Vermeeren MA, Ommen VV, Wildberger JE. Prophylactic hydration to protect renal function from intravascular iodinated contrast material in patients at high risk of contrast-induced nephropathy (AMACING): a prospective, randomised, phase 3, controlled, open-label, non-inferiority trial. Lancet. 2017 Apr 1;389(10076):1312-1322. doi: 10.1016/S0140-6736(17)30057-0. Epub 2017 Feb 21. PMID 28233565
- [Background] Centraal BegeleidingsOrgaan (CBO). CBO richtlijnen contrast. 2007 Available from: www.cbo.nl/product/richtlijnen/folder20021023121843/rl_jodium_2007
- [Background] Veligheids Management Systeem. VMS veiligheidsprogramma. Voorkomen van nierinsufficiëntie bij intravasculair gebruik van jodiumhoudende contrastmiddelen. September 2009. 2009 [cited; Available from: http:/www.vmszorg.nl/10- Themas/Nierinsufficientie/Praktijkgids-Nierinsufficientie
- [Derived] Nijssen EC, Nelemans PJ, Rennenberg RJ, van der Molen AJ, van Ommen GV, Wildberger JE. Impact on clinical practice of updated guidelines on iodinated contrast material: CINART. Eur Radiol. 2020 Jul;30(7):4005-4013. doi: 10.1007/s00330-020-06719-7. Epub 2020 Feb 27. PMID 32107605